CLINICAL TRIAL: NCT01776983
Title: Skin Aging in Renal Transplant Patients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2008SIA01
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Photosensitivity Disorders
MeSH Terms: conditions — Photosensitivity Disorders

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Photosensitivity under the influence of immunocomp — Siascopy measurement of reflected light

SUMMARY:
Determination of collagen, pigment and haemoglobin content of sun exposed and sun protected skin by Siascopy. Immunocompromised patients (for more than seven years) compared to immunocompetent patients.

* Trial in the field of transplantation / xenotransplantation

DETAILED DESCRIPTION:
Determination of collagen, pigment and haemoglobin content of sun exposed and sun protected skin by Siascopy. Immunocompromised patients (for more than seven years) compared to immunocompetent patients.

ELIGIBILITY:
Inclusion criteria:

* Renal transplant recipients transplanted more than seven years ago and immunocompetent probands of the same age.

Exclusion criteria:

* Refusal of informed consent, physical or psychological inability to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: individuals between 18 and 90 years of age
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
skin aging defined by melanin, collagen and hemoglobin content | One Time measurement at the one and only time point of inclusion and measurement
  there is only one time point for measurement, there is no "time frame", just one single measurement per patient at the one and only visit

CONTACTS AND LOCATIONS:
Overall Officials: Günther Hofbauer, MD, Principal Investigator — University Hospital Zurich, Department of Dermatology
Locations (1):
- University Hospital Zurich, Department of Dermatology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Result] Stimpfle DW, Serra AL, Wuthrich RP, French LE, Braun RP, Hofbauer GF. Spectophotometric intracutaneous analysis: an investigation on photodamaged skin of immunocompromised patients. J Eur Acad Dermatol Venereol. 2015 Jun;29(6):1141-7. doi: 10.1111/jdv.12771. Epub 2014 Oct 13. PMID 25307045